CLINICAL TRIAL: NCT04961723
Title: Randomized Control Trial of Home-based Hepatitis C Self-testing in Key Populations in Georgia
Brief Title: HCV Self-testing in Georgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: National Center for Disease control and Public Health (Other Government); Batumi Imedi Harm Reduction Site (Unknown); Equality Movement (Unknown); Center for Information and Counseling on Reproductive Health - Tanadgoma (Other); Tbilisi New Way Harm Reduction Site (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: HC022
Record Dates: First submitted 2021-06-19; First posted 2021-07-14 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C; Diagnostic Self Evaluation
Keywords: People who inject drugs (PWID); Men who have sex with men (MSM); Linkage to care; Online self-test distribution; self-test
MeSH Terms: conditions — Hepatitis C; Homosexuality

STUDY DESIGN:
Intervention Model Description: 5 arm randomized control trial evaluating models of care by population group. For MSM group 3 arms; a postal delivery model of HCV antibody self-test, a peer delivery model of HCV antibody self-test compared the standard or care (participant going to clinic for HCV antibody RDT).
  For PWID 2 arms; a peer delivery model of HCV antibody self-test compared the standard or care (participant going to clinic for HCV antibody RDT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MSM Postal delivery (Experimental): Participants who identify primarily as MSM will receive a home delivered HCV self-test kit in non-identifiable packaging. The kit will include the test, instructions for use (IFU), and information about additional supporting materials, such as access to live chat and a call center for questions about testing
  Interventions: Diagnostic Test: (OraQuick® HCV Self-Test
- MSM Peer delivery (Experimental): Participants who identify primarily as MSM will schedule a peer delivery of the HCV self-test kit and IFU. The peer will provide basic information about the test, what to do if the test is reactive, and how to access to live chat and a call center for questions about testing
  Interventions: Diagnostic Test: (OraQuick® HCV Self-Test
- MSM control (No Intervention): Participants who identify primarily as MSM will receive information about standard of care HCV antibody testing available at local testing sites in their community. Participants will also have access to live chat and a call center for questions about HCV testing
- PWID peer delivery (Experimental): Participants who identify primarily as PWID will schedule a peer delivery of the HCV self-test kit and IFU. The peer will provide basic information about the test, what to do if the test is reactive, and how to access to live chat and a call center for questions about testing
  Interventions: Diagnostic Test: (OraQuick® HCV Self-Test
- PWID control (No Intervention): Participants who identify primarily as PWID will receive information about standard of care HCV antibody testing available at local testing sites in their community. Participants will also have access to live chat and a call center for questions about HCV testing

INTERVENTIONS:
Diagnostic Test: (OraQuick® HCV Self-Test — The OraQuick® HCV Self-Test is a lateral flow rapid diagnostic that can detect anti-HCV antibodies in oral fluid. Instructions for Use (IFU) for OraQuick® HCV Rapid Antibody Self-Test have been developed in Georgian for the previous 2 studies conducted in Georgia using the OraQuick® HCV Rapid Antibody Self-Test. The IFU has been optimized taking in the feedback on the IFU resulting from the aforementioned studies. As this HCV test is not approved for self-test use in Georgia, all tests will be labelled as Research Use Only (RUO) and test results will not be used for patient management.
  Arms: MSM Peer delivery; MSM Postal delivery; PWID peer delivery

SUMMARY:
Self-testing with easy-to-use rapid diagnostic tests has been successfully used for diseases such as HIV. The availability of self-testing has been shown to increase testing rates and testing acceptability in diverse populations around the world, in large part due to its convenience and privacy advantages.7 Self-testing has also been effectively used to reach key populations who may not be covered by traditional healthcare programs, such as persons who inject drugs (PWID) and men who have sex with men (MSM). In Georgia, HIV self-testing has been offered to MSM through an online platform promoting their uptake.11-12 In the present study aims to evaluate the acceptability and impact of using an online platform to enable home delivery of HCV self-testing in Georgia for PWID and MSM.

DETAILED DESCRIPTION:
Georgia, a middle-income country with an estimated population of 3.7 million people, is among the world's highest-burden countries for HCV, with an estimated sero-prevalence of 7.7% in the general population and a higher burden of disease in high-risk populations such as persons who inject drugs. In 2015, Georgia embarked on an elimination program for HCV which includes the expansion of HCV testing, linkage to care, and treatment.

The country made a substantial progress in HCV testing, linkage to care and treatment during the last five years, but the gap still remains that needs to be addressed through testing of different screening modalities to reach marginalized groups of the population.

Self-testing with easy-to-use rapid diagnostic tests has been successfully used for diseases such as HIV. The availability of self-testing has been shown to increase testing rates and testing acceptability in diverse populations around the world, in large part due to its convenience and privacy advantages. The present study aims to evaluate the acceptability and impact of an online program enabling home delivery of HCV self-testing (HCVST) for people who inject drugs (PWID) and men who have sex with men (MSM) in Georgia.

The National Centres for Disease Control (NCDC) and FIND, in conjunction with the Georgian national HCV elimination program, Batumi Imedi, Equality Movement, Tanadgoma, and Tbilisi New Way are evaluating HCV self-testing as a way to expand outreach, improve HCV testing rates, and increase linkage to care among HCV-infected PWID and MSM. The ability to utilize an existing online platform promoting HIV self-testing, selftest.ge, will enable the study to examine how offering HCV self-testing may help Georgia reach its goal of nationwide elimination of HCV

The study aims to describe the acceptability and impact of an online platform offering home delivery of HCV self-tests to PWID and MSM. Since HCV self-tests detect the presence of antibodies to HCV, indicating exposure to HCV, any individual reporting a positive HCV self-test will be referred to HCV RNA confirmatory testing in order to identify active HCV infection. Those confirmed to have active HCV infection with a positive HCV RNA test will be linked to HCV treatment and care. Rates of testing and linkage to care will be measured, along with knowledge, attitudes, and practices around HCV testing and care

This is a randomized controlled trial comparing an online platform providing home-delivery of HCV self-tests to referral to standard of care community-based HCV testing sites in PWID and MSM in Georgia.

Study participants will be recruited through an existing HIV self-testing program using an online platform to promote the study. Interested participants will sign up to be contacted for study eligibility screening and consent. All study participants will complete a baseline survey collecting demographics and knowledge and attitudes towards HCV testing.

Randomization will be done among participants who primarily identify as MSM (arm 1, 2 and 3) and separately among participant who primarily identify as PWID

* Arm 1: MSM postal delivery Participants who identify primarily as MSM will receive a home delivered HCV self-test kit in non-identifiable packaging. The kit will include the test, instructions for use (IFU), and information about additional supporting materials, such as access to live chat and a call center for questions about testing
* Arm 2: MSM peer delivery Participants who identify primarily as MSM will schedule a peer delivery of the HCV self-test kit and IFU. The peer will provide basic information about the test, what to do if the test is reactive, and how to access to live chat and a call center for questions about testing
* Arm 3: MSM control Participants who identify primarily as MSM will receive information about standard of care HCV antibody testing available at local testing sites in their community. Participants will also have access to live chat and a call center for questions about HCV testing
* Arm 4: PWID peer delivery Participants who identify primarily as PWID will schedule a peer delivery of the HCV self-test kit and IFU. The peer will provide basic information about the test, what to do if the test is reactive, and how to access to live chat and a call center for questions about testing
* Arm 5: PWID control Participants who identify primarily as PWID will receive information about standard of care HCV antibody testing available at local testing sites in their community. Participants will also have access to live chat and a call center for questions about HCV testing All participants will be sent a telephone reminder Follow-up survey #1 which includes the opportunity to upload any testing result approximately 2-4 weeks after enrolment. A second Follow-up survey will be sent after the closure of the first survey. Up to 3 reminders may be sent for each survey if a survey has not been completed. Participants will receive 10 GEL phone credit (~3 USD) for completion of the first follow up questionnaire to enter test result and an additional 10 GEL for completion of the follow-up survey.

Any participants who report HCV antibody positive result through the study will be contacted by the project staff and offered confirmatory testing and appropriate linkage to care through the national HCV program. For all arms study staff will contact to the participants who report HCV antibody positive result via the online platform and will provide information about the next steps for diagnostic and treatment, information about the treatment facilities. Those participants will be contacted again after 6 weeks and will be asked if they received the next HCV care.

The HCV test used in the intervention group is an oral fluid test (OraQuick® HCV Self-Test). Although use as a self-test is still research use only, it has been validated by the manufacturer for self-testing. The test has also already been CE marked and WHO pre-qualified as an in vitro diagnostic for professional use by healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able and eligible to access services on selftest.ge
* Self-identify as a PWID and or MSM
* Living in Batumi or Tbilisi
* Able to understand the scope of the study and provide informed consent through online platform.
* Able to read and understand Georgian
* Unknown HCV serology status (i.e., never tested for HCV or tested HCV ab- in a most recent test performed no later than 6 months before enrolment)

Exclusion Criteria:

* Self-reported previously confirmed positive HCV status (either Ab or RNA)
* Un-eligible for Georgian National Hepatitis Elimination program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — for MSM arms participant eligibility is based on if a person self-identifies as a men who has sex with men
Enrollment: 1250 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of HCV self-testing home delivery on HCV antibody testing rates in PWID and MSM | 2 weeks to 2 months after enrollment
  The number of participants who report completing the HCV antibody testing in the intervention group vs the control group
To assess the impact of HCV self-testing home delivery on HCV antibody testing rates in PWID and MSM | 2 weeks to 2 months after enrollment
  To assess that the proportion of participants who report completing the HCV antibody testing in the intervention group is superior to that of the participants in the control group by a margin of 20%.

SECONDARY OUTCOMES:
To assess the impact of HCV self-testing on the number of HCV antibody positive individuals who are aware of their status | 2 weeks to 2 months after enrollment
  Number of HCV antibody positive participants made aware of their status in the intervention vs control group
To assess the impact of HCV self-testing on linkage and completion of HCV RNA confirmatory testing in HCV antibody positive individuals | 2 weeks to end of study
  2.2 The number of HCV antibody positive participants who are referred to and complete HCV RNA confirmatory testing in the intervention vs control group
To assess the impact of HCV self-testing on treatment initiation in HCV RNA positive individuals eligible to start treatment | 2 weeks to end of study
  2.3 The number of HCV RNA positive participants who start treatment in the intervention vs control group
To assess the acceptability of HCV self-testing at baseline and after study participation. | 2 weeks to 3 months after enrollment
  2.4 Analysis of survey responses using proportions and means. The responses to the questionnaire at baseline and after study participation will be compared to assess if there are changes in acceptability of HCV self-testing
To assess the cost of HCV self-testing | entire duration of study, estimated 6 months
  Cost per test completed, cost per person diagnosed (serology, RNA) in the intervention vs control groups. The costs of each step on the testing pathway will be combined to determine the overall cost per person diagnosed with HCV viremia

CONTACTS AND LOCATIONS:
Overall Officials: Ketevan Stvilia, Principal Investigator — National Center for Disease Control and Public Health, Georgia
Locations (6):
- Georgia (6):
  - Center for Information and Counselling on Reproductive Health-Tanadgoma, Batumi
  - Equality Movement, Batumi
  - Imedi Harm Reduction Site, Batumi
  - Center for Information and Counselling on Reproductive Health-Tanadgoma, Tbilisi
  - Equality Movement, Tbilisi
  - Tbilisi New Way Harm Reduction Site, Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shilton S, Stvilia K, Japaridze M, Tsereteli N, Usharidze D, Phevadze S, Jghenti M, Mozalevskis A, Markby J, Luhmann N, Johnson C, Nabeta P, Ongarello S, Reipold EI, Gamkrelidze A. Home-based hepatitis C self-testing in people who inject drugs and men who have sex with men in Georgia: a protocol for a randomised controlled trial. BMJ Open. 2022 Sep 8;12(9):e056243. doi: 10.1136/bmjopen-2021-056243. PMID 36691209